CLINICAL TRIAL: NCT00448656
Title: Treatment of Atrial Fibrillation by Minimal Invasive Epicardial Pulmonary Vein Isolation: The ABOLISH-AF Study
Brief Title: Treatment of Atrial Fibrillation by Minimal Invasive Surgery
Acronym: ABOLISH-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, I.C. Van Gelder, Prof.dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: p06.0550l
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; epicardial ablation pulmonary veins; video assisted thoracic surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ablation of pulmonary veins by video assisted thoracic surgery — epicardial ablation using HIFU
  Other Names: Epicor

SUMMARY:
The purpose of this study is to determine the feasability of a new epicardial and minimal invasive ablation technique of the left atrium isolating the pulmonary veins for prevention of atrial fibrillation recurrences in patients with antiarrhythmic drug refractory lone atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation is a major health problem.Despite adequate treatment of underlying heart disease, rhythm control is unsuccessful in almost half of patients, also in patients with lone atrial fibrillation.If patients remain highly symptomatic, a non-pharmacological approach may be considered including pulmonary vein isolation and Cox maze III surgery. Maze III surgery has high succes rates, however it includes major cardiac surgery with substantial risk of complications. New surgical strategies for symptomatic lone atrial fibrillation focus on minimal invasive off-pump procedures omitting cardiopulmonary bypass (and thus lowering the complication rate), while taking advantage of an easier approach to the ablation site and a shorter procedure time. Epicardial surgical ablation isolating pulmonary veins by high intensity focused ultrasound performed off-pump by Video Assisted Thoracic Surgery (VATS)may be a promising treatment option. In this pilot study, we aim to study the feasibility of this new surgical ablation approach in patients with lone atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic lone paroxysmal or persistent atrial fibrillation, which either convert spontaneously or can be terminated with antiarrhythmic drugs or by an electrical cardioversion.
2. The patient had a least one episode of persistent atrial fibrillation or three episodes of paroxysmal atrial fibrillation during the last three months.
3. Duration present episode persistent atrial fibrillation less then one year.
4. The patient has been treated with at least two different antiarrhythmic drugs (class I-IV) of which at least one belongs to class I or III.
5. The patient will sign and date the written informed consent prior to study participation.

Exclusion Criteria:

1. Age <18 and >76 years.
2. Contraindications for oral anticoagulation.
3. Signs of sick sinus syndrome or AV conduction disturbances (i.e. symptomatic bradycardia or asystole > 3 seconds or escape rate < 40 beats per minute in awake symptom-free patients).
4. Permanent atrial fibrillation defined as atrial fibrillation continuously present and not convertible to sinus rhythm by an electrical cardioversion or antiarrhythmic drugs.
5. Previous transvenous pulmonary vein isolation, Maze surgery, or other cardiac surgery.
6. Heart failure defined as NYHA class III-IV heart failure.
7. Previously implanted intracardiac device or has current or foreseen pacemaker, internal cardioverter defibrillator (ICD) and/ or cardiac resynchronization therapy.
8. Clinically relevant valvular heart disease.
9. Coronary artery disease or an old myocardial infarction
10. Acute or chronic infection.
11. Untreated clinical hypo- or hyperthyroidism or < 3 months euthyroidism.
12. Uncontrolled hypertension, defined as a systolic blood pressure > 160 mm Hg and/or a diastolic blood pressure > 95 mm Hg (anti-hypertensive treatment is allowed).
13. The patient has a concurrent medical condition (i.e. alcohol or drug abuse or a severe progressive extracardiac disease) or is unlikely to comply with the protocol.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
sinus rhythm at end of follow-up (6 months) | 6 months

SECONDARY OUTCOMES:
absence of permanent atrial fibrillation at end of follow-up | 6 months
absence of any symptomatic atrial fibrillation | 6 months
atrial volume and contraction at end of follow-up | 6 months
left ventricular diameters and function at end of follow-up | 6 months
thromboembolism | 6 months
pulmonary vein stenosis | 6 months
immediate postoperative complications (and related sequelae) | directly post-operative
surgical procedure time and total epicardial ablation time | directly post-operative
any pacemaker implantation | 6 months
mortality | 6 months
bleeding | 6 months
hospitalization for heart failure | 6 months
antiarrhythmic drugs during follow-up | 6 months
electrical cardioversions during follow-up | 6 months
re-ablations | 6 months
syncope | 6 months
quality of life and specific arrhythmia symptoms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C. Vam Gelder, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Klinkenberg TJ, Ahmed S, Ten Hagen A, Wiesfeld AC, Tan ES, Zijlstra F, Van Gelder IC. Feasibility and outcome of epicardial pulmonary vein isolation for lone atrial fibrillation using minimal invasive surgery and high intensity focused ultrasound. Europace. 2009 Dec;11(12):1624-31. doi: 10.1093/europace/eup299. Epub 2009 Oct 6. PMID 19812047